CLINICAL TRIAL: NCT02425228
Title: Paired CAP: Prospective Assessment of Image Registration for the Diagnosis of Prostate Cancer
Brief Title: Prospective Assessment of Image Registration for the Diagnosis of Prostate Cancer
Acronym: Paired Cap
Status: Completed | Type: Observational
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 14-000990; JCCCID481 (Other: Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2015-03-23; First posted 2015-04-23 (Estimated); Last update posted 2020-07-24 (Actual); Status verified 2019-05

CONDITIONS: Elevated PSA; Prostate Cancer
Keywords: targeted biopsy; conventional biopsy; cognitive biopsy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Targeted biopsy — conventional/systematic biopsy, targeted fusion biopsy and cognitive biopsy

SUMMARY:
This is a pilot study to determine cancer detection rate of conventional/systematic versus targeted biopsy methods in diagnosis of potentially lethal prostate cancer. This is a diagnostic trial using each patient as his own control.

DETAILED DESCRIPTION:
Each biopsy session would be preceded by mpMRI, which would be delineated and assigned a degree of suspicion by a radiologist (see above).The PI-RADS scoring system will be used to assign a degree of suspicion to regions of interest within the prostate. A second reader will independently score the RSI on a Likert scale, blinded to the other MRI data. The regions of interest will be delineated using software developed by Eigen in collaboration with a study co-author (D.M.), now commercially available and in use by the UCLA team for the past 2 years (ProFuse, Eigen).The RSI data will be integrated with the standard mpMRI data and any change in scoring or presence of additional lesions, determined by RSI, will be quantified. For men with a MR-visible target of PI-RADS score 3 or more, irrespective of RSI score, the biopsy session would then proceed in an ordered routine, as follows:

1. Conventional ultrasound-guided 12-core systematic biopsy would be performed first. This portion will be performed without operator knowledge of the MRI report, i.e., the urologist will be blinded to possible tumor location and use the method in standard practice throughout the U.S. for many years.
2. Next a targeted biopsy would be performed using visual guidance (cognitive fusion), under the supervision of a radiologist specializing in prostate MRI. The radiologist will be in the biopsy suite and help the urologist direct needle at location of region of interest in the prostate seen on MRI. Three directed biopsy cores will be obtained.
3. Third, a targeted biopsy using Artemis device fusion of MRI and ultrasound images would be performed. The prostate will be scanned and the MRI region of interest (target) brought into the 3D model via device fusion. Targeted biopsy will be performed by taking three cores of tissue from the target area, visualized as a 3D region in the fusion device.

Biopsy sites to be dictated by geometric guides (12 point pattern vs visual direction of radiologist vs fusion target), not chosen arbitrarily.

The above biopsy schema will not require any more procedure time or samples taken than fusion biopsy as performed under IRB approval at our institution for the last five years. Additional cores will be required for the visual biopsy method, but no biopsy cores will be obtained from secondary targets. Most patients exhibit secondary targets. An analysis of data from past 2 years demonstrated that the chance of a secondary target showing significant cancer, not present in a primary target, is less than 1%. Therefore, secondary targets will not be sampled, as cores are instead taken from primary targets using the two methods. In 200 men undergoing initial biopsy, an average of 17 +/- 3 S.D. cores/patient has been obtained. In the present proposal, 18 cores will be taken. Thus, the number of cores/patient in this trial will not substantially exceed the number that has been routinely taken in our practice in the past.

A sampling method of three directed cores per target was chosen as a compromise between what is clinically feasible and a statistical ideal of taking additional cores for significant cancer detection in lower grade targets.

The cognitive biopsy will require approximately 90 seconds of additional time, but this added time will be more than compensated by the reduced time obtained from excluding secondary targets. The overall biopsy schema should require no more (and probably less) than the 15-20 minutes/procedure as in the past. Biopsies will be performed by an experienced team, which has been working together since 2009.

ELIGIBILITY:
Inclusion Criteria:

* Men undergoing a first-time prostate biopsy driven by PSA elevation to rule out cancer.
* PSA 2.5 - 20 ng/mL
* Prostate volume 20 - 100 cc
* No prior ablation or TURP
* Able to tolerate MRI
* T1c suspect
* Signed informed consent

Exclusion Criteria:

* Any prior prostate biopsy
* Active bleeding disorder or concurrent use of coumadin or any other anticoagulant, unless anticoagulation can be temporarily stopped for at least 7 days before and 7 days after the biopsy
* Any prostate ablative procedure, including transurethral resection, photovaporization, or electrovaporization
* Any contraindication to MRI (contrast allergy, severe claustrophobia, MRI-incompatible prosthesis) ,
* Palpable prostate mass lesion (i.e., Stage >T1c suspected)
* Any condition that would preclude the subject from getting the required biopsy as stated in the protocol

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Men with targetable lesion on MRI, undergoing a first-time prostate biopsy driven by PSA elevation to rule out cancer.
  We choose to study men undergoing first-time biopsy, since the great challenge with prostate biopsy today is to establish a correct diagnosis initially. The study sample is kept uniform by excluding men with prior negative biopsies and men enrolled in the Active Surveillance program. Men without a targetable lesion and men with a PI-RADS <2 lesion currently undergo a mapping biopsy under an existing IRB approval; data collection on these men would continue in parallel, but would not be part of this targeting study
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2014-12-04 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2018-12-18 (Actual)

PRIMARY OUTCOMES:
Detection of clinically significant cancer | one DAY
  Patient participation is only confined to the biopsy visit.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UCLA, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California